CLINICAL TRIAL: NCT00566540
Title: Intensification Regimen for Previously Untreated, Resectable, Advanced Squamous Cell Carcinoma of the Oral Cavity, Oropharynx, and Hypopharynx: Incorporation of Intensity Modulated Radiotherapy and Submandibular Gland Transfer to Minimize Treatment Morbidity; Correlative Imaging/Molecular Markers.
Brief Title: Ph 2 Intensification Regimen for Previously Untreated, Resectable, Advanced Squamous Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems with study
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Enver Ozer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06026; NCI-2011-02687 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Paclitaxel; Radiotherapy, Intensity-Modulated; Radiotherapy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (neoadjuvant, adjuvant chemotherapy and radiation) (Experimental): PREOPERATIVE:Patients receive cisplatin IV over 2 hours three times weekly in week 1 once daily(QD),5 days a week, in weeks 1-2.
  SURGERY:Patients undergo triple endoscopy and biopsy with submandibular gland transfer in week 3.
  INTRAOPERATIVE: Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation.
  POSTOPERATIVE: Patients receive paclitaxel IV over 3 hours in weeks 7-10 and cisplatin IV over 1-2 hours three times weekly in weeks 7 and 10. Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation QD, 5 days a week, in weeks 7-10.
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Radiation: Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation; Procedure: Triple endoscopy and biopsy

INTERVENTIONS:
Drug: Cisplatin — Patients will receive Cisplatin (30 mg/m2 i.v.) daily x 3 days in week 1.
  Other Names: Platinol-®AQ; cis-DDP; cis-Diamminedichloroplatinum; cis-Platinum II; DDP
Drug: Paclitaxel — Patients will receive Paclitaxel (45 mg/m2i.v.) infusion over 3 hours during weeks 7,8,9,10
  Other Names: Taxol®
Radiation: Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation — Patients will receive Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation to tumor and involved regional nodes 20Gy over 10 daily (M-F) treatments (2 Gy Fractions with 6 millivolts photons)week 1 and 2.
  Other Names: radiation therapy; EBT; IMRT
Procedure: Triple endoscopy and biopsy — Resection of the primary tumor: Patients must have surgery performed according to the following surgical guidelines. The extent of the surgical resection will be dictated by the extent of the tumor at the time of initial evaluation. The primary lesion must be widely excised using accepted criteria for adequate excision depending on the region involved. All patients will undergo percutaneous endoscopic gastrostomy tube placement at the time of endoscopy and biopsies.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving cisplatin and paclitaxel together with radiation therapy and surgery works in treating patients with advanced cancer of the oral cavity, oropharynx, or hypopharynx that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of a new intensification regimen comprising cisplatin and paclitaxel in combination with radiotherapy and surgery in patients with resectable advanced squamous cell carcinoma of the oral cavity, oropharynx, or hypopharynx.

Secondary

* Assess the disease-free interval and failure sites in patients treated with this regimen.
* Correlate molecular markers with treatment outcome in these patients.
* Correlate quality of life with treatment outcome in these patients.
* Determine the frequency and severity of toxicities of this regimen in these patients.
* Evaluate treatment completion in these patients.

OUTLINE:

* Preoperative therapy (weeks 1 and 2): Patients receive cisplatin IV over 2 hours on days 1-3. Patients also undergo intensity-modulated external beam radiotherapy once daily on days 1-5 and 8-12.
* Surgery (week 3): Patients undergo surgical resection of the primary tumor (with or without neck dissection) and intraoperative boost radiotherapy.
* Postoperative therapy (weeks 7-10): Patients receive cisplatin IV over 2 hours on days 1-3 and 22-24 and paclitaxel IV over 3 hours on days 1, 8, 15, and 22. Patients also undergo intensity-modulated external beam radiotherapy on days 1-5, 8-12, 15-19, and 22-26.

Patients undergo blood and tissue sample collection at baseline, in weeks 3, 7-10, and 14, and then periodically thereafter for biomarker correlative studies.

Quality of life is assessed at baseline, at 3, 6, and 12 months after completion of treatment, and then annually thereafter.

After completion of study treatment, patients are followed every 2 months for 1 year and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky Performance Index ≥60%
* Patients must be over the age of 18.
* Patients must have a life expectancy of at least 6 months.
* Women of childbearing age must have a negative serum pregnancy test and agree to use an effective method of contraceptive.
* Patients with a cardiac history should be cleared with a medical internist. In general, patients with a history of prior bradyarrythmias, atrioventricular (AV) conduction defects or marginal cardiac function will be eligible.
* Patients must have resectable stage III, stage IVA, stage IVB (without distant metastases) squamous cell carcinoma of the oral cavity, oropharynx, or hypopharynx. Hypopharyngeal carcinomas may also be stage II.
* Patients must not have had prior chemotherapy or radiotherapy (to the primary site or nodes).
* Patients may not be planning to receive while on study concomitant immunotherapy or hormonal therapy, except oral contraceptives or hormone replacement therapy.
* Patients must have adequate hepatic function documented by a normal serum bilirubin 0- 1.5mg/L and serum transaminases < 4 x upper limit.
* Patients must have adequate renal function documented by a serum creatinine not above upper institutional normal limits and/or 24 hour OR calculated creatinine clearance >60 ml/min. using the following formula:

  (140-age) x Wt (kg) x .85 (if Estimated Creatinine Clearance = 72 x Creatinine (mg/dl) female)
* Patients must have adequate bone marrow function documented by platelet count ≥ 100,000 and absolute neutrophil count ≥ 2,000.
* Patients will have surgery according to Section 5.3. Operative and pathology reports must be sufficiently detailed to confirm that surgery was done according to the guidelines.
* Patients must be examined by a multi-modality team (consisting of a head and neck surgeon, medical oncologist, and radiation oncologist) prior to entry on study.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Distant metastases.
* Prior malignancy, except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years.
* Any condition that would be considered a contraindication for fluid challenge.
* Pregnant or lactating women may not participate.
* History of demyelinating neurological disorder, such as multiple sclerosis
* History of pancytopenia or aplastic anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12-11 (Actual); Primary Completion 2010-02-25 (Actual); Study Completion 2010-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enver Ozer, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation): PREOPERATIVE:Patients receive cisplatin IV over 2 hours 3 times weekly in week 1 once daily(QD),5 days a week, in weeks 1-2.
  SURGERY:Patients undergo triple endoscopy and biopsy with submandibular gland transfer in week 3.
  INTRAOPERATIVE: Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation.
  POSTOPERATIVE: Patients receive paclitaxel IV over 3 hours in weeks 7-10 and cisplatin IV over 1-2 hours three times weekly in weeks 7 and 10. Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation QD, 5 days a week, in weeks 7-10.
  Cisplatin: Patients will receive Cisplatin (30 mg/m2 i.v.) daily x 3 days in week 1.
  Paclitaxel: Patients will receive Paclitaxel (45 mg/m2i.v.) infusion over 3 hours during weeks 7,8,9,10 Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation: Patients will receive Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation to tumor and involved regional nod
Period: Overall Study
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation): PREOPERATIVE:Patients receive cisplatin IV over 2 hours three times weekly in week 1 once daily(QD),5 days a week, in weeks 1-2.
  SURGERY:Patients undergo triple endoscopy and biopsy with submandibular gland transfer in week 3.
  INTRAOPERATIVE: Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation.
  POSTOPERATIVE: Patients receive paclitaxel IV over 3 hours in weeks 7-10 and cisplatin IV over 1-2 hours three times weekly in weeks 7 and 10. Patients also undergo Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation QD, 5 days a week, in weeks 7-10.
  Cisplatin: Patients will receive Cisplatin (30 mg/m2 i.v.) daily x 3 days in week 1.
  Paclitaxel: Patients will receive Paclitaxel (45 mg/m2i.v.) infusion over 3 hours during weeks 7,8,9,10 Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation: Patients will receive Intensity-Modulated Radiation Therapy (IMRT) External Beam Radiation to tumor and involved regional nod
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 63 [49 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Treatment
Description: Determine the feasibility of a new intensification regimen for previously untreated resectable advanced stage head and neck cancer that incorporates Cisplatin, Paclitaxel combined with surgery, submandibular gland transfer and radiation therapy
Time Frame: Up to one year
Population: The data was not collected or analyzed due to discontinuation of study in early stages.
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease-free Interval and Failure Sites
Description: Assess disease-free interval and failure sites of a new treatment regimen.
Time Frame: Up to one year
Population: The data was not collected or analyzed due to discontinuation of study in early stages.
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Quality of Life With Treatment Outcome
Description: Assess quality of life with treatment outcome will be obtained at baseline (prior to treatment) and at 6 months post treatment and one year post-treatment follow-ups.
Time Frame: Up to one year
Population: The data analysis was unable to be completed due to discontinuation of study in early stages
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: Determine the frequency and severity of toxicities of the intensification regimen. Patients will be evaluated for local and systemic toxicity/morbidity from treatment regimen.
Time Frame: Up to one year
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 11
percentage of patients
  Leukocytes | 9
  Rash | 9
  Colitis | 9
  Dehydration | 18
  Diarrhea | 9
  Vomiting | 9
  Hemorrhage, Upper Respiratory | 9
  Infection with normal ANC | 9
  Edema | 9

5. Secondary Outcome: Treatment Completion
Description: Patients are to be seen at Ohio State Medical center for a physical exam every 2 months for the first year.
Time Frame: up to one year
Population: The data analysis was unable to be completed due to discontinuation of study in early stages
Measure: Number; unit: patients
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 11
patients | 7

6. Other Pre Specified Outcome: Correlation of Molecular Markers With Treatment Outcome
Description: Evaluate potential correlative molecular markers with treatment outcome
Time Frame: Up to week 14
Population: The data was not collected or analyzed due to discontinuation of study in early stages.
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events were graded using the NCI Common Toxicity Criteria version 3.0.
Arm/Group | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation)
All-Cause Mortality (participants affected / at risk) | 2/11
Serious Adverse Events (participants affected / at risk) | 11/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation) (N=11)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Neck NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Neoadjuvant, Adjuvant Chemotherapy and Radiation) (N=11)
Extremity pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Edema-limb (General disorders) | 4 (4)
Oral cavity pain (Gastrointestinal disorders) | 10 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Salivary gland changes (Gastrointestinal disorders) | 4 (4)
Mucositis/stomatitis (Gastrointestinal disorders) | 10 (10) — oral cavity
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Fatigue (General disorders) | 10 (10)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 10 (10)
Neutrophils/granulocytes/ANC (Blood and lymphatic system disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8)
Throat/pharynx, larynx pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Weight loss (Investigations) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 7 (7) — sensory
Vomiting (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 8 (8)
ALT (serum glutamic pyruvic transaminase) (Investigations) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 9 (9)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 9 (9)
Face pain (General disorders) | 4 (4)
Edema-head and neck (General disorders) | 9 (9)
Infection (Infections and infestations) | 7 (7) — Infection with normal ANC or Grade 1 or 2 neutrophils - Oral cavity-gums (gingivitis)

LIMITATIONS AND CAVEATS:
The study was stopped in the early stages and no data analysis was completed and results produced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes